CLINICAL TRIAL: NCT02686983
Title: Greater Occipital Nerve Blockade for the Treatment of Chronic Migraine: a Randomized, Double- Blind, Placebo-controlled Study
Brief Title: GON-block in Chronic Migraine: a Randomized, Double- Blind, Placebo-controlled Study
Acronym: DHC-GON-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jakob Møller Hansen, MD. (Other)
Responsible Party: Sponsor-Investigator, Jakob Møller Hansen, MD., MD, PhD, Danish Headache Center
Organization: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: DHC-GON-1
Record Dates: First submitted 2016-02-12; First posted 2016-02-22 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — Betamethasone; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Betamethasone and local anesthetic.
  Interventions: Drug: Betamethasone and local anesthetic
- Placebo (Placebo Comparator): Saline with local anesthetic.
  Interventions: Drug: Betamethasone and local anesthetic

INTERVENTIONS:
Drug: Betamethasone and local anesthetic — Infiltration of the greater occipital nerve .
  Other Names: GON block

SUMMARY:
Infiltration of the greater occipital nerve (GON) with local anaesthetics and corticosteroids is a treatment option for cluster headache. Corticosteroids may be helpful in reducing the pain intensity and frequency in chronic migrtaine. This RCT is set up to assess efficacy and safety of sub-occipital steroid injections with local anesthetic in patients with chronic migraine.

DETAILED DESCRIPTION:
Infiltration of the greater occipital nerve (GON) with local anaesthetics and corticosteroids is a treatment option for cluster headache. In general, there is a marked paucity of evidence concerning GON blocks in migraine. Corticosteroids may be helpful in reducing the pain intensity and frequency in these patients. This is an RCT to assess efficacy and safety of sub-occipital steroid injections with local anesthetic in patients with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine

Exclusion Criteria:

* Medication overuse headache

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of migraine days | 8 weeks
  Number of days fulfilling the ICHD criteria for migraine

SECONDARY OUTCOMES:
Number of days with severe headache days | 8 weeks
  Number of days with severe headache days
Medication use | 8 weeks
  use of medication recorded during the 8 weeks
Responder rate | 8 weeks
  number of patients with more than 50% reduction in migraine
Number of migraine attacks | 8 weeks
  Number of attacks fulfilling the ICHD criteria for migraine

CONTACTS AND LOCATIONS:
Overall Officials: Jakob M Hansen, MD, PhD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, University of Copenhagen, Faculty of Health Sciences, Department of Neurology, Glostrup Hospital, Glostrup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided